CLINICAL TRIAL: NCT04741295
Title: To Study the Effect of Low Molecular Weight Heparin on the Adenomyosis Patients'Outcome of in Vitro Fertilization-embryo Transplantation
Brief Title: Low Molecular Weight Heparin on the Adenomyosis Patients'IVF-ET Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Professor, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SZ-2021-ADE1
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Adenomyosis; Assisted Reproductive Technology
MeSH Terms: conditions — Adenomyosis | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Adenomyosis patients in control group have normal luteal progesterone support.
- Low molecular weight heparin Group (Experimental): Adenomyosis patients in Low molecular weight heparin group have Low molecular weight heparin in addition to normal luteal progesterone support.
  Interventions: Drug: Low molecular weight heparin

INTERVENTIONS:
Drug: Low molecular weight heparin — Patients with adenomyosis were treated with low molecular weight heparin after frozen embryo transfer in addition to routine luteal support.
  Arms: Low molecular weight heparin Group

SUMMARY:
In assisted reproductive technology, adenomyosis patients are characterized by lower clinical pregnancy rate, lower implantation rate and higher abortion rate. The purpose of this study is to explore whether low molecular weight heparin can reduce the abortion rate of adenomyosis patients in frozen thawed embryo transfer cycles.

ELIGIBILITY:
Inclusion Criteria:

1. The basal serum level of FSH was less than 10 IU / L
2. Diagnosed with adenomyosis by ultrasound
3. The first frozen thawed embryo transfer cycle, by hormone replacement protocol
4. Transfer at least one high quality frozen embryo;
5. Patients agreed to use low molecular weight heparin after FET, and they were able to sign informed consent in person.

Exclusion Criteria:

1. With abnormal karyotype;
2. Accompanied with other uterine diseases: intrauterine adhesion, intramural myoma, moderate to severe endometriosis, congenital uterine malformation, endometrial tuberculosis, thin endometrium < 8mm on the day of transformation, etc;
3. PCOS, RIF patients;
4. There are indications of conventional anticoagulation or antiplatelet therapy, such as antiphospholipid syndrome, autoimmune diseases, coagulation dysfunction, etc;
5. There were contraindications to hormone replacement therapy and low molecular weight heparin;
6. Participating in other clinical studies;
7. Unable to follow-up

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Early spontaneous abortion rate | Within three months after frozen embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No